CLINICAL TRIAL: NCT04960345
Title: Comparison of Accuracy and Clinical Outcomes Between Brainlab Knee 3 Computer-assisted Navigation Systems and Conventional Instruments in TKA: a Prospective Cohort Study
Brief Title: Comparison Between Brainlab Knee 3 Computer-assisted Navigation Systems and Conventional Instruments in TKA: a Prospective Cohort Study.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: navigation68480
Record Dates: First submitted 2021-07-04; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Total Knee Arthroplasty
Keywords: Total knee arthroplasty; Lower limb alignment; Navigation; Functional outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- The traditional group: The traditional group underwent prosthesis placement using traditional intramedullary positioning method.
- The navigation group: The navigation group performed surgery using the Brainlab Knee 3 navigation system.Informed consent was signed after grouping.
  Interventions: Device: Brainlab Knee 3

INTERVENTIONS:
Device: Brainlab Knee 3 — Brainlab knee 3 navigation system is a kind of imageless computer-assisted navigation system.
  Other Names: Brainlab knee 3 navigation system
  Groups: The navigation group

SUMMARY:
This is a a prospective cohort study. According to the inclusion criteria, volunteers were recruited from patients undergoing total knee arthroplasty. The patients are devided into two groups: the conventional TKA,the computer-assisted surgery(CAS) using Brainlab Knee 3 system.The differences of postoperative alignment,operative time,blood loss will be studied between the two groups.Clinical and functional evaluation using the scoring system of HSS(Hospital for Special Surgery) score, Western Ontario and McMaster University osteoarthritis index (WOMAC), Forgotten joint score(FJS-12) will be compared between the 2 groups,after surgery, and at the follow-up of 3 months、6 months and 12 months.

DETAILED DESCRIPTION:
According to the inclusion criteria, patients receiving primary total knee arthroplasty were recruited and divided into two groups after doctor-patient joint decision: the traditional group underwent prosthesis placement using traditional intramedullary positioning method;The navigation group performed surgery using the Brainlab Knee 3 navigation system.Informed consent was signed after grouping. All patients were operated by the same knee prosthesis system. Both groups underwent the same procedures such as the installation of the soft tissue adjustment, prosthesis placement, wound closure and so on.All patients were given the same perioperative treatment, such as hemostasis, anti-infection and analgesia, and routine postoperative rehabilitation exercises. The full length anteroposterior and lateral radiographs of both lower extremities in weight-bearing position were taken preoperatively and one week postoperatively.The differences of postoperative alignment,operative time,blood loss will be studied between the two groups.Clinical and functional evaluation using the scoring system of HSS(Hospital for Special Surgery) score, Western Ontario and McMaster University osteoarthritis index (WOMAC), Forgotten joint score(FJS-12) will be compared between the 2 groups,after surgery, and at the follow-up of 3 months、6 months and 12 months.

ELIGIBILITY:
Inclusion criteria:

1. Patients with knee osteoarthritis who underwent primary TKA;
2. Informed consent has been signed and medical records are complete;
3. No severe varus or valgus deformity of the knee (< 20°).

Exclusion criteria:

1. Patients undergoing revision knee replacement;
2. patients with rheumatoid arthritis and secondary knee osteoarthritis;
3. Patients with severe valgus deformity(≥ 20°);
4. Taking anticoagulant drugs for a long time in the past, or suffering from the following diseases: Renal insufficiency, liver insufficiency, severe heart disease (or coronary stent implantation within the last 12 months), severe respiratory disease, history of deep vein thrombosis in the lower extremities or a high risk of thrombosis (hereditary/acquired thrombosis), coagulation dysfunction, stroke, and malignancy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with knee osteoarthritis who underwent primary TKA
Sampling Method: Non-Probability Sample
Enrollment: 188 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
lower limb alignment | Within 1 week after surgery
  knee-ankle angle (HKA) and components placement using coronal femoral-component angle (CFA) and coronal tibia- component angle (CTA)、sagittal femoral-component angle (SFA) and sagittal tibia-component angle（STA）.

SECONDARY OUTCOMES:
Operation time | Immediately after surgery
  Time from skin incision to wound closure.
Blood loss | 3 days after surgery
  Postoperative drainage volume refers to the drainage volume of the affected knee within 24 hours after the end of surgery, accurate to ml.Gross linear equation was used to calculate the total blood loss and latent blood loss at 3 days after surgery.
the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 3 months、6 months and 12 months after surgery
  The WOMAC is a self administered questionnaire to assess joint function and quality of life for patients with osteoarthritis; it consists of 24 items: pain (5 items), stiffness (2 items), and physical function (17 items). The higher the total score, the worse the patient's pain, stiffness, and functional limitations. The WOMAC is validated for various languages, including Chinese.
HSS(Hospital for Special Surgery) score | 6 months and 12 months after surgery
  HSS(hospital for special surgery) score HSS(hospital for special surgery) score to evaluate patients postoperative knee joint function. With a total of 100, it has 7 subscales: 1.Pain 0~30; 2. Function 0~22; 3. Mobility 0~18; 4. Flexion deformity 0~10; 6. Stability 0~10; 7. Deduction Item. For each scale, a higher value represents a better outcome. The sum of the subscales is the total score.
Forgotten Joint Score-12 (FJS-12) | 6 months and 12 months after surgery
  The FJS-12 is a PROM for patients who have undergone a TKA; it introduces the concept of a "forgotten" joint as the ideal objective to pursue in prosthetic surgery. It is composed of 12 items, measuring the patient's ability to forget the presence of an artificial joint in their daily life. For each item, there is a five-points Likert scale response. The raw results are converted to a 0-100 points scale. Highest score corresponds to good outcome with the patient not aware about the presence of the prosthesis. In the case of more than 4 answers are missing, the score should not be used .